CLINICAL TRIAL: NCT03036241
Title: Drug-eluting Balloon vs. Conventional Balloon in the Treatment of (re)Stenosis - a Randomized Prospective Study (Dialysis Fistulae)
Brief Title: Drug-eluting Balloon vs. Conventional Balloon in the Treatment of (re)Stenosis (Dialysis Fistulae)
Acronym: DRECOREST2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, Professor of Vascular Surgery, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRECOREST2 - 23rd Jan 2013
Record Dates: First submitted 2017-01-19; First posted 2017-01-30 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Vascular Access Complication; Restenosis, Vascular Graft; Dialysis Related Complications
Keywords: drug-eluting balloon,; target lesion revascularization (TLR); restenosis
MeSH Terms: conditions — Graft Occlusion, Vascular | interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-eluting balloon (Experimental)
  Interventions: Device: Angioplasty with drug-eluting balloon
- Conventional angioplasty (Active Comparator)
  Interventions: Device: Conventional angioplasty

INTERVENTIONS:
Device: Conventional angioplasty — Angioplasty with conventional balloon
  Other Names: PTA
  Arms: Conventional angioplasty
Device: Angioplasty with drug-eluting balloon — Angioplasty with drug-eluting balloon
  Other Names: DEB
  Arms: Drug-eluting balloon

SUMMARY:
The purpose of this study is to determine whether the use of drug-eluting balloons is effective in the treatment of (re)stenosis in dialysis fistulae.

DETAILED DESCRIPTION:
Drug-eluting devices have proved beneficial in the treatment of stenosis in native coronary and lower limb arteries. Stenosis and restenosis is a known problem in dialysis fistulae and drug-eluting devices might be beneficial in this field as well.

In the procedure a conventional balloon is passed through the stenosis which is then dilated. After this patients are randomized before a second dilatation with either a conventional balloon or a drug-coated balloon.

The stenosis is evaluated preoperatively and followed up by means of ultrasound by a vascular technician. Follow-up will end at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Any dialysis access w/ native vessels warranting intervention

Exclusion Criteria:

* Previous PTA with drug-eluting balloon, thrombolysis, coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01-23 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
TLR | 12 months
  Target lesion revascularization, ie. re-intervention to the same lesion
Occlusion of access | 12 months
  Any loss of dialysis access due to thrombosis

SECONDARY OUTCOMES:
Primary assisted patency | 12 months
  Patency after endovascular reintervention due to restenosis or thrombosis
Death | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maarit Venermo, Prof, Principal Investigator — Helsinki University Hospital, dept of vascular surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjorkman P, Weselius EM, Kokkonen T, Rauta V, Alback A, Venermo M. Drug-Coated Versus Plain Balloon Angioplasty In Arteriovenous Fistulas: A Randomized, Controlled Study With 1-Year Follow-Up (The Drecorest Ii-Study). Scand J Surg. 2019 Mar;108(1):61-66. doi: 10.1177/1457496918798206. Epub 2018 Sep 5. PMID 30182815